CLINICAL TRIAL: NCT03516097
Title: TeenPower: e-Empowering Teenagers to Prevent Obesity
Acronym: TeenPower
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Instituto Politécnico de Castelo Branco (Other); Polytechnic University of Santarém (Other); Município de Leiria (Unknown)
Responsible Party: Principal Investigator, Pedro Sousa, Prof., Instituto Politécnico de Leiria
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POCI-01-0145-FEDER-23557
Record Dates: First submitted 2018-04-14; First posted 2018-05-04 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Adolescent Obesity; Empowerment; ICT
MeSH Terms: conditions — Pediatric Obesity; Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A (Experimental): Structured school based intervention + mobile app usage
  Interventions: Behavioral: Structured school based intervention; Device: mobile app usage
- Experimental Group B (Experimental): mobile app usage
  Interventions: Device: mobile app usage
- Control Group (Active Comparator): Structured school based intervention
  Interventions: Behavioral: Structured school based intervention

INTERVENTIONS:
Behavioral: Structured school based intervention — Intervention includes behavioral, nutritional and physical activity counselling (online and face-to-face psycho-educative sessions).
  Arms: Control Group; Experimental Group A
Device: mobile app usage — The e-therapeutic platform and mobile app (TeenPower) includes educational resources, self-monitoring, social support, interactive training modules and motivational tools. In addition to the case manager, the program will also have the direct support of an interdisciplinary team (nurse, nutritionist, exercise physiologist, psychologist among others).
  Arms: Experimental Group A; Experimental Group B

SUMMARY:
Transdisciplinary practice-based action research project that aims to develop innovative cognitive-behavioral interventions to empower adolescents, through increased and interactive contact between adolescent and multidisciplinary healthcare team. Project born from the discussion with trans-territorial stakeholders (health professionals and school communities), in the absence of an integrated, creative and dynamic strategy of overweight prevention and promotion of salutogenic behaviors in adolescents.

The polytechnics of Leiria, Santarém and Castelo Branco are co-promotors of this project, as well as Município de Leiria (City Council), key partners in the development and implementation of the intervention program. It is expected the partnership with ARS-Centro.

The main goal is the development, implementation and evaluation of a program for the promotion of healthy behaviors and prevention of obesity in adolescence, based on e-therapy and sustained by the case management methodology.

DETAILED DESCRIPTION:
Transdisciplinary practice-based action research project that aims to develop innovative interventions to promote healthy behaviors. Project called from a territorial issue, identified and discussed with local stakeholders (health professionals and school community), in the absence of an integrated, creative and dynamic strategy of overweight prevention and promotion of salutogenic behaviors in adolescents.

Adolescent obesity has reached epidemic proportions, being urgent to find effective prevention strategies and adequate resources that induce change at the individual, family and community level. The core components of classic prevention programs have been unable to obtain the desired adherence. The solution may involve a more extensive and frequent contact with the healthcare team and the use of alternative communication channels and interacting/dynamic technologies with adolescents.

Given the research team's experience in developing innovative products and healthcare technological solutions, this need was faced as an opportunity to network and explore synergies between territorial partners. The polytechnics of Leiria (IPL), Santarém (IPS) and Castelo Branco (IPCB) are co-promotors of this project, as well as the Município de Leiria (City Council). It is also expected the partnership with the local primary healthcare stakeholders (Administração Regional de Saúde do Centro: ARS-C), key partners in the development phase and in the implementation of the intervention program. An agile product development process will be adopted, an iterative and incremental approach for planning and implementing, in an intense and permanent dialogue with healthcare professionals, and adolescents throughout the platform and the mobile app development process.

The main goal is the development, implementation and evaluation of a program for the promotion of healthy behaviors and prevention of obesity in adolescence, based on e-therapy and sustained by the case management methodology. The project is directed to the cognitive-behavioral empowerment of adolescents, through increased and interactive contact between adolescents and multidisciplinary healthcare team. The use of Information and Communication Technologies (ICT) in the intervention can optimize resources and maximize impact, as a complement to conventional approaches, The project includes the development of three complementary studies: (S1) evaluation of adolescents' health status and cognitive-behavioral indicators, (S2) usability evaluation of the TeenPower platform and mobile app (S3) implementation and adherence evaluation to the TeenPower intervention program.

The positive evaluation of the intervention program will stimulate the inclusion of ICT in the promotion of salutogenic behaviors and overweight prevention, creating technological interfaces that will allow customizing the intervention parameters and facilitating the monitoring and tracking.

ELIGIBILITY:
Inclusion Criteria:

* school groups of Leiria, Santarém and Castelo Branco, aged between 12 and 16, with easy access to internet and smartphone/tablet

Exclusion Criteria:

* language or cognitive limitations

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline BMI at 3 months | Month 3
  Body Mass Index
Change from baseline Physical activity at 3 months | Month 3
  Questionnaire "Quantification de l'Activité Physique en Altitude Chez les Enfants"
Change from baseline Nutrition at 3 months | Month 3
  Questionnaire on adolescent food choices
Change from baseline Adolescent Lifestyle at 3 months | Month 3
  Adolescent Lifestyle Profile Questionnaire
App usability | Month 3
  usability questionnaire
User experience | Month 3
  User experience questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Politécnico de Leiria, Leiria, Portugal

IPD SHARING:
Plan to Share IPD: Undecided